CLINICAL TRIAL: NCT01693172
Title: Effect of an Early Mobilization Program After Surgery on Functional Recovery and Clinical Complications in Patients Undergoing Major Cancer Surgey : a Randomized Controlled Trial
Brief Title: Effect of an Early Mobilization Program on Outcomes After Major Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, Elisangela P M de Almeida, MD, Principal Investigator, Instituto do Cancer do Estado de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 118/12
Record Dates: First submitted 2012-09-07; First posted 2012-09-26 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Neoplasm
Keywords: exercise; neoplasm
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- early postoperative mobilization (Active Comparator): Early postoperative supervised aerobic exercise, resistance and flexibility training
  Interventions: Behavioral: Early mobilization program
- Standard (No Intervention): Standard rehabilitation care

INTERVENTIONS:
Behavioral: Early mobilization program — Early postoperative supervised aerobic exercise, resistance and flexibility training
  Arms: early postoperative mobilization

SUMMARY:
The aim of this study is to evaluate the effect of an early postoperative physical rehabilitation program on the functional capacity and incidence of postoperative complications in patients undergoing major elective surgery for treatment of a neoplasm

ELIGIBILITY:
Inclusion Criteria:

* Patients who will be submitted to major surgery for cancer treatment.
* Age ≥ 18 years
* Reading and signing the informed consent

Exclusion Criteria:

Acute myocardial infarction (within the last 30 days)

* Unstable Angina
* Cardiac arrhythmia uncontrolled
* symptomatic severe aortic stenosis
* Congestive heart failure NYHA III or IV
* infarction or acute pulmonary thromboembolism
* pericarditis or myocarditis
* Acute Endocarditis
* Acute aortic dissection
* Active infection
* Acute renal failure
* Thyrotoxicosis
* Refusal to participate in the study
* Inability to ambulate independently and / or inability to exercises
* Presence of bone metastasis
* musculoskeletal and neurological conditions that preclude the achievement of an exercise program designed for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Ability to walk three meters or crossing a room without assistence | at 5 days after surgery or at hospital discharge

SECONDARY OUTCOMES:
fatigue | at 5 and 30 days after surgery
  We will assess the level of fatigue through the Piper fatigue scale
quality of life | at 5, 30, 180 and 365 days after surgery
length of hospital stay | at hospital discharge
recurrence of cancer | at 180 days after surgery
hospital costs | at 180 days after surgery
post operatorative complications | at 30 days after surgery
  Clavien classification

CONTACTS AND LOCATIONS:
Overall Officials: Ludhmila A Hajjar, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Instituto do Câncer do Estado de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] de Almeida EPM, de Almeida JP, Landoni G, Galas FRBG, Fukushima JT, Fominskiy E, de Brito CMM, Cavichio LBL, de Almeida LAA, Ribeiro U Jr, Osawa EA, Diz MP, Cecatto RB, Battistella LR, Hajjar LA. Early mobilization programme improves functional capacity after major abdominal cancer surgery: a randomized controlled trial. Br J Anaesth. 2017 Nov 1;119(5):900-907. doi: 10.1093/bja/aex250. PMID 28981596